CLINICAL TRIAL: NCT01684956
Title: Pharmacokinetic Comparison of Intradermal Versus Sub-cutaneous Insulin and Glucagon Delivery in Volunteers With Type 1 Diabetes
Brief Title: Pharmacokinetic Comparison of Intradermal Versus Sub-cutaneous Insulin and Glucagon Delivery in Type 1 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012P001098
Record Dates: First submitted 2012-08-23; First posted 2012-09-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Type 1 Diabetes
Keywords: intradermal; pharmacokinetics; microneedle; insulin; glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Injections, Intradermal; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal first (Experimental): Intradermal injection experiment first, followed by subcutaneous injection experiment
  Interventions: Procedure: Intradermal injection; Procedure: Subcutaneous injection
- Subcutaneous first (Experimental): Subcutaneous injection experiment first, followed by intradermal injection experiment
  Interventions: Procedure: Intradermal injection; Procedure: Subcutaneous injection

INTERVENTIONS:
Procedure: Intradermal injection
Procedure: Subcutaneous injection

SUMMARY:
The investigators are doing this research study to find out if the type of needle used to administer them affects the speed with which insulin and glucagon get into the blood. The investigators will compare a traditional insulin needle to an injection device, called the MicronJet, that uses microneedles to deliver medication into the top layer of your skin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older with clinical type 1 diabetes for at least one year
* Diabetes managed using an insulin infusion pump and rapid- or very-rapid-acting insulins including insulin aspart (Novolog), insulin lispro (Humalog), and insulin glulisine (Apidra).
* Ability to consume a sufficient amount of carbohydrates over 2-3 hours to cover 5 units of rapid acting insulin
* Stimulated C-peptide <0.1 nmol/L at 90 minutes after liquid mixed meal tolerance test.

Exclusion Criteria:

* Unable to provide informed consent
* Unable to comply with study procedures
* Current participation in another diabetes-related clinical trial other than one that is primarily observational in nature. Potential subjects enrolled in trails of passive monitoring equipment, such as continuous glucose monitors (CGMs), are not excluded
* Inadequate venous access as determined by study nurse or physician at time of screening
* Pregnancy
* Hemoglobin less than 13.5 for men and less than 12 for women
* History of pheochromocytoma (fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor to include episodic or treatment refractory hypertension defined as requiring 4 or more medications to achieve normotension, paroxysms of tachycardia, pallor, or headache, or personal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease)
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting
* History of adrenal disease or tumor
* Hypertension (blood pressure > 160/100 mm/Hg at screening or day of study visit
* History of allergy to aspirin or any history of aspirin intolerance, including Reye's syndrome, or gastric ulcer or bleeding associated with salicylates.
* Blood dyscrasia or bleeding diathesis, such as hemophilia, Von Willebrand's disorder, and idiopathic thrombocytopenic purpura (ITP)
* Peptic Ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Aggregate mean difference in tmax between the delivery methods (the insulin and glucagon data will be evaluated separately) | 1 day

SECONDARY OUTCOMES:
Aggregate mean difference in t1/2max between the methods | 1 day visit
Aggregate mean difference in Cmax between the methods | 1 day
Aggregate mean difference in area under the curve (AUC) between methods | 1 day
AUC of 0-1 hour (and by subtraction hours 1-5) | 1 day
AUC of 0-2 hours (and by subtraction hours 2-5) | 1 day
Time to 50% of Total AUC (or said another way, time to 50% exposure) | 1 day
Fraction of subjects with difference in tmax between the methods of > 25% | 1 day
Fraction of "dry" injections with no reflux of fluid from the injection site | 1 day
Difference in mean visual analog pain score between the two methods | 1 day
Difference in mean visual analog pain score between insulin and glucagon with subcutaneous injection | 1 day
Difference in mean visual analog pain score between insulin and glucagon with intradermal injection | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States